CLINICAL TRIAL: NCT04548141
Title: Simplification de l'évaluation de l'Activité PHysique Par Interrogatoire Rapide
Brief Title: Quick Questionnaire to Evaluate Physical Activity
Acronym: SAPHIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Principal Investigator, DENISE JOLIVOT, Doctor, University Hospital, Angers
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SAPHIR
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Sedentary Behavior
Keywords: Physical activity; Questionnaire
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Self completion of questionnaire in the waiting room
Masking Description: Anonymous completion of questionnaire
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active adults (Experimental): Adults coming for a visit for sports activity participation and submitted the SAPHIR questionnaire
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Scoring of the IPAQ is performed according to references. Scoring of the SAPHIR has been submitted for copyright protection (involves a series of 23 additions)

SUMMARY:
The purpose of this study is to test and validate a new questionnaire (SAPHIR) in order to get an evaluation of patients physical activity.

DETAILED DESCRIPTION:
Two questionnaires the SAPHIR and the "International Physical Activity Questionnaire" (IPAQ) are submitted (self completion) to patients referred for consultation.

Retrival of physical activity data on podometer if available

ELIGIBILITY:
Inclusion Criteria:

* French Native language
* Covered by the French social care system
* Be referred for a consultation to the Sports Medicine Service of Angers Hospital or to the CRSS of Angers

Exclusion Criteria:

* Person opposed to participating in the research
* Person unable to understand the objectives of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

PRIMARY OUTCOMES:
Proportion of questionnaires with errors after self completion | 1 day
  Estimation of the percentage of errors with 90% confidence interval Comparison of the two percentages

SECONDARY OUTCOMES:
Facility of the filling of the questionnaires | 1 day
  Ease of use évaluation for the patient using Likert scale (from "Totally agree" to "not agree at all" in 5 grades)
Correlation of the SAPHIR questionnaire to the IPAQ questionnaire | 1 day
  Correlation coefficient with the IPAQ questionnaire
Correlation of the SAPHIR questionnaire to the number of weekly steps for patients who have a pedometer available | 1 day
  The correlation coefficient with the number of steps will be studied

CONTACTS AND LOCATIONS:
Overall Officials: Pierre ABRAHAM, Principal Investigator — University and Hospital in Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: No